CLINICAL TRIAL: NCT00752050
Title: A Phase 3, Multi-Center Trial to Demonstrate the Safety and Efficacy of Repeat Treatment With PurTox® for the Treatment of Glabellar Rhytides ("Frown Lines")
Brief Title: Safety and Efficacy Study of Repeat Treatment With PurTox® Botulinum Toxin Type A for Frown Lines Between the Eyebrows
Acronym: PT-03b
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Mentor Worldwide, LLC (Industry)
Collaborators: Synteract, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: PT-03b
Record Dates: First submitted 2008-09-11; First posted 2008-09-15 (Estimated); Last update posted 2011-09-12 (Estimated); Status verified 2011-09

CONDITIONS: Glabellar Rhytides; Frown Lines Between the Eyebrows
Keywords: Botulinum Toxin Type A; Botulinum Toxin; Glabellar Rhytides; Rhytides; Frown Lines; Neuromuscular Agents; Neurotoxin; Forehead; Eyebrow; Wrinkle
MeSH Terms: interventions — Botulinum Toxins, Type A; Botulinum Toxins; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Mentor Purified Toxin Botulinum Toxin Type A - Part II ONLY. (Part I is Single Group and all participants receive active drug and are not randomized)
  Interventions: Drug: Mentor Purified Toxin Botulinum Toxin Type A
- 2 (Placebo Comparator): Preservative-free Saline - Part II ONLY. (Part I is Single Group and all participants receive active drug and are not randomized)
  Interventions: Drug: Preservative-free Saline

INTERVENTIONS:
Drug: Mentor Purified Toxin Botulinum Toxin Type A — For Part II, subjects in this arm will receive five 0.1 mL intramuscular injections at the Day 0 Treatment Visit: two in each corrugator and one in the procerus muscle. The total treatment dose (sum of the five injections) to be administered will be 30 U of the Active Comparator Mentor Purified Toxin.
  Other Names: Botulinum Toxin Type A; Botulinum Toxin
  Arms: 1
Drug: Preservative-free Saline — For Part II, subjects in this arm will receive five 0.1 mL intramuscular injections at the Day 0 Treatment Visit: two in each corrugator and one in the procerus muscle. The total treatment dose (sum of the five injections) to be administered will be 0.5 mL of the placebo (preservative-free saline).
  Other Names: Saline
  Arms: 2

SUMMARY:
The overall purpose of this study is to evaluate the safety and effectiveness of repeat treatment of an intramuscular dose of Mentor Purified Toxin for the reduction of frown lines, compared with placebo.

DETAILED DESCRIPTION:
The purpose of this a randomized withdrawal Phase III, multi-center research study is to evaluate the safety and effectiveness of repeat treatment with an intramuscular dose of Mentor Purified Toxin in the reduction of glabellar rhytides (frown lines). Approximately 700 subjects will be enrolled at approximately 12 clinical sites in the U.S.A.

Effectiveness will be determined by the degree of frown line reduction, during maximum forced frown and at rest (neutral expression):

* as assessed live by the study doctor,
* as assessed live by the subject, and;
* as assessed by an independent reviewer based on subject photographs

Frown lines are graded on level of severity based on this scale:

Severity

* Minimal (0)
* Mild (1)
* Moderate (2)
* Severe (3)

There are two parts to this study. In the first part, all study participants will receive treatment with an intramuscular injection of 30 Units of Mentor Purified Toxin on two separate occasions (Cycles 1 and 2) no more than 6 months apart. In the second part of the study (Cycle 3), subjects will be randomly assigned to receive either intramuscular injections of 30 Units of Mentor Purified Toxin or placebo (preservative-free saline) and subjects will be followed for 1 month (3:1, PurTox : placebo).

Each subject will receive five intramuscular injections for a total of 0.5 mL of study drug in the glabellar area, during each treatment visit. Participation takes place over a maximum of 14 months, including Part 1 (Cycle 1 and 2) and Part 2 (Cycle 3). The number of clinic visits will vary from person to person depending upon the subject's response to the study drug, but will range from approximately 9 to 19 clinic visits. There will also be up to 4 telephone follow-up contacts.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects who are 18 years of age or older (subjects should have an interest in the effacement of glabellar rhytides) with or without previous botulinum Toxin Type A exposure;
2. In good physical and mental health as determined by the investigator based on medical history, physical examination, and/or clinical laboratory tests;
3. Noticeable presence of the glabellar rhytides for a period of 6 months or longer;
4. Score at least a 2 (moderate severity) at baseline screening on the investigator's and subject's assessments (reference photographs provided) at forced frown; and
5. Capable of understanding and complying with the protocol and must have signed the informed consent document prior to performance of any study-related procedures.

Exclusion Criteria:

1. A history of psychiatric problems that, in the investigator's opinion, is severe enough potentially to interfere with subject outcomes;
2. A history of autoimmune disease, that, in the opinion of the investigator, might interfere with subject outcomes (e.g., osteoarthritis is not considered an exclusion criteria; however, subjects with dermatomyositis are not permitted to participate in this study);
3. A history or presence of clinically significant cardiovascular, respiratory, hepatic/biliary, renal, gastrointestinal, endocrinological, or neurological disorders constituting a possible risk factor that, in the investigator's opinion, is severe enough potentially to interfere with subject outcomes;
4. Inability to substantially efface glabellar lines by manually spreading skin apart;
5. Eyelid ptosis;
6. Myasthenia gravis (from medical history or diseases of neurotransmission);
7. Current history of facial nerve paralysis;
8. Concurrent dermatologic disease of the face in the glabellar area that is deemed by the investigator to make the subject an inappropriate candidate for the study;
9. Recent flu-like syndrome that, in the investigator's opinion, is severe enough potentially to interfere with subject outcomes;
10. Neuromuscular disorder that, in the investigator's opinion, is severe enough potentially to interfere with subject outcomes;
11. Active multisystems disease that, in the investigator's opinion, might influence the outcome measures or the safety of the subject;
12. Has any condition(s) that in the investigator's opinion would a) warrant exclusion from the study, or b) prevent the subject from completing the study;
13. Currently receiving aminoglycoside antibiotic therapy, curare-like drugs, quinidine, succinylcholine, polymyxins, anticholinesterases, magnesium sulfate, or lincosamides;
14. Has taken any investigational drug during the 30 days prior to screening visit;
15. Have had Botulinum Toxin treatments to the glabellar and/or forehead area during the 6 months prior to screening visit;
16. Have had dermal filler treatment to glabellar area during the 6 months prior to screening visit;
17. Female subjects who are pregnant or lactating. Female subjects who are of childbearing potential must have negative urine pregnancy test results prior to enrollment into the study. Such subjects, including peri-menopausal women who have had a menstrual period within one year, must be using appropriate birth control (see protocol/informed consent for description);
18. Unwilling or unable to comply with the protocol or to cooperate fully with the investigator and site personnel; and
19. Unable to understand verbal and/or written English or any other language in which a certified translation of the informed consent document is available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 699 (Actual)
Dates: Start 2007-11; Primary Completion 2009-02 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
Change in assessments of severity of glabellar rhytide by the investigator and the subject at maximum frown as a single composite effectiveness endpoint. | Day 30 post randomization
Measurement of the incidences of treatment-emergent adverse events, serious treatment-emergent adverse events, treatment-emergent laboratory abnormalities, and vital signs. | Throughout

SECONDARY OUTCOMES:
Change in assessments of severity of glabellar rhytide by the investigator and the subject at maximum frown. | Day 30 post-injection
Change in assessments of severity of glabellar rhytide by the investigator and the subject at rest. | Day 30 post randomization
Change in assessments of severity of glabellar rhytide by independent reviewers based on the photographs of the subject's glabellar lines at maximum frown. | Baseline and Day 30 post randomization

CONTACTS AND LOCATIONS:
Overall Officials: Corey Maas, MD, Study Director
Locations (1):
- Mentor Wordwide, LLC, Santa Barbara, California, United States